CLINICAL TRIAL: NCT03519711
Title: A Phase 1/2, Open-Label, Randomized Parallel Arm, Intra-patient Dose Escalation Study to Evaluate the Safety, Pharmacokinetics and Preliminary Efficacy of CNSA-001(Sepiapterin) in Primary Tetrahydrobiopterin Deficient Patients With Hyperphenylalaninemia
Brief Title: A Study of PTC923 (CNSA-001) in Primary Tetrahydrobiopterin (BH4) Deficient Participants With Hyperphenylalaninemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBD-001
Record Dates: First submitted 2018-04-11; First posted 2018-05-09 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2022-05

CONDITIONS: BH4 Deficiency; Hyperphenylalaninemia
MeSH Terms: conditions — Phenylketonurias | interventions — sepiapterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: PTC923 2.5 and 10 mg/kg/day (Experimental): Participants will receive PTC923 suspension 2.5 milligrams (mg)/kilogram (kg)/day (dose divided in 2 for twice daily administration) orally for 7 days in Period 1, undergo a 3 (±1) day washout period, then escalate to a dose of 10 mg/kg/day (dose divided in 2 for twice daily administration) administered orally for 7 days in Period 2 (14 days total treatment).
  Interventions: Drug: PTC923
- Cohort 2: PTC923 5 and 20 mg/kg/day (Experimental): Participants will receive PTC923 suspension 5 mg/kg/day (dose divided in 2 for twice daily administration) orally for 7 days in Period 1, undergo a 3 (±1) day washout period, then escalate to a dose of 20 mg/kg/day (dose divided in 2 for twice daily administration) administered orally for 7 days in Period 2 (14 days total treatment).
  Interventions: Drug: PTC923

INTERVENTIONS:
Drug: PTC923 — PTC923 will be administered per dose and schedule specified in arm description.
  Other Names: CNSA-001, Sepiapterin

SUMMARY:
This study has been designed to demonstrate the safety, pharmacokinetics (PK) and preliminary efficacy of PTC923 (CNSA-001) in reducing blood phenylalanine concentrations in participants with hyperphenylalaninemia due to primary BH4 deficiency (PBD).

DETAILED DESCRIPTION:
BH4 is an essential cofactor for phenylalanine hydroxylase, tyrosine hydroxylase, tryptophan hydroxylase, fatty acid glycerylether oxygenase, and nitric oxide (NO) synthase. The PBD is caused by deficiency of GTP cyclohydrolase I (GTP-CH), 6-pyruvoyl-tetrahydropterin synthase (PTPS), or sepiapterin reductase (SR) that impairs the biosynthesis of BH4 or by defects in BH4 recycling (pterin-4a-carbinolamine dehydratase [PCD] or dihydropteridine reductase [DHPR] deficiency).

Participants will be randomized into one of 2 cohorts, with each cohort assessing 2 dose levels of PTC923 via intra-participant escalation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 years old and above and 12 months old and above for the remaining participants (age reduction pending analysis of safety, PK, and response, in the adult participant(s) by the Data Safety Monitoring Board (DSMB) and Food and Drug Administration [FDA])
* Confirmed diagnosis of PBD as evidenced by medical history of biallelic pathogenic mutations in PTPS or recessive GTP-CH genes, abnormal enzymatic activity of the PTPS or GTP-CH enzymes, or a cerebrospinal fluid (CSF) biochemical profile indicative of PTPS or GTP-CH deficiencies
* Informed consent and assent (if necessary) with parental consent
* Females must be either postmenopausal for ≥1 year, or surgically sterile (tubal ligation, hysterectomy, or bilateral oophorectomy) for at least 6 months or, if of childbearing potential and not abstinent, willing to use at least 2 of the following highly effective methods of contraception (including adolescents 12 to 18 years old) from screening through 30 days after the last dose of study drug:

  * Hormonal contraception (stable dose for 3 months)
  * Intrauterine device/intrauterine hormone-releasing system
  * Barrier contraceptive method (diaphragm, cervical cap, contraceptive sponge, condom) with spermicidal foam/gel/cream/suppository Males and females who are abstinent will not be required to use a second contraceptive method unless they become sexually active.
* Males with female partners of childbearing potential must agree to use barrier contraceptive (that is, condom) with spermicidal foam from screening through 90 days after the last dose of study drug. Males must also refrain from sperm donations during this time period.
* Females with a negative pregnancy test at screening and on Day 1 prior to dosing
* Creatinine clearance (CrCl) >90 milliliters (mL)/minute (min) as estimated using the Cockcroft-Gault equation (≥18 years) or Schwartz-Lyon equation (≥12 months <18 years)
* The participant is clinically stable on therapy for management of their signs and symptoms of PBD as determined by the investigator.
* The participant is willing and able to comply with the protocol.
* No tobacco use (for example; cigarettes, e-cigarettes, cigars, smokeless tobacco) for 2 weeks prior to the screening visit and willingness to abstain from these products through the last dose of study drug

Exclusion Criteria:

* PBD caused by biallelic pathogenic mutations in PCD, SR, DHPR, or single dominant mutations in GTP-CH
* Significant chronic medical illness other than PBD, as determined by the investigator
* Gastrointestinal disease (such as irritable bowel syndrome, inflammatory bowel disease, chronic gastritis, peptic ulcer disease, etc.) that could affect the absorption of study drug
* History of gastric surgery, including Roux-en-Y gastric bypass surgery or an antrectomy with vagotomy, or gastrectomy
* Inability to tolerate oral medication
* History of allergies or adverse reactions to BH4 or related compounds, or any excipients in the study drug formulation
* Any clinically significant medical or psychiatric condition or medical history, that in the opinion of the investigator, would interfere with the participant's ability to participate in the study or increase the risk of participation for that participant
* Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) laboratory values >2 * the upper limit of normal (ULN)
* Any other clinically significant laboratory abnormality unrelated to PBD at the screening visit or prior to the administration of the first dose of study drug, as determined by the investigator
* Clinically significant cardiac arrhythmia at screening or prior to the first dose of study drug
* QTcF (QT with Fridericia's correction) ≥460 milliseconds (msec) in males and ≥480 msec in females (based on the mean of triplicate measurements taken at screening)
* Resting heart rate ≤40 or ≥110 beats/minute (bpm) for ages 12 and older, ≥130 bpm for ages 3 to 12, ≥150 bpm for ages 1 to 2 years, or resting blood pressure <85/40 millimeters of mercury (mmHg) or >150/90 mmHg at screening or prior to the first administration of study drug
* Current participation in any other investigational drug study or participation within 30 days prior to screening
* History of alcohol or drug abuse within last 6 months prior to screening or current evidence of substance dependence as determined by the investigator
* Currently taking an antifolate including, but not limited to, methotrexate, pemetrexed, or trimetrexate
* A female who is nursing or who is pregnant or planning to become pregnant.
* The participant, in the opinion of the investigator, is unwilling or unable to adhere to the requirements of the study.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Smith, PharmD, Study Director — Censa Pharmaceuticals
Locations (4):
- United States (4):
  - University of Minnesota, Minneapolis, Minnesota
  - UT Southwestern, Dallas, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Marshfield Clinic, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: PTC923 2.5 and 10 mg/kg/Day: Participants received PTC923 (CNSA-001) suspension 2.5 milligrams (mg)/kilogram (kg)/day (dose divided in 2 for twice daily administration) orally for 7 days in Period 1, underwent a 3 (±1) day washout period, then escalated to a dose of 10 mg/kg/day (dose divided in 2 for twice daily administration) administered orally for 7 days in Period 2 (14 days total treatment).
- Cohort 2: PTC923 5 and 20 mg/kg/Day: Participants received PTC923 suspension 5 mg/kg/day (dose divided in 2 for twice daily administration) orally for 7 days in Period 1, underwent a 3 (±1) day washout period, then escalated to a dose of 20 mg/kg/day (dose divided in 2 for twice daily administration) administered orally for 7 days in Period 2 (14 days total treatment).
Period: Treatment Period 1 (7 Days)
Arm/Group | Cohort 1: PTC923 2.5 and 10 mg/kg/Day | Cohort 2: PTC923 5 and 20 mg/kg/Day
Started | 4 | 4
Received at Least 1 Dose of Study Drug | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Treatment Period 2 (7 Days)
Arm/Group | Cohort 1: PTC923 2.5 and 10 mg/kg/Day | Cohort 2: PTC923 5 and 20 mg/kg/Day
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population included all randomized participants who received any amount of study drug.
Groups:
- Cohort 1: PTC923 2.5 and 10 mg/kg/Day: Participants received PTC923 suspension 2.5 mg/kg/day (dose divided in 2 for twice daily administration) orally for 7 days in Period 1, underwent a 3 (±1) day washout period, then escalated to a dose of 10 mg/kg/day (dose divided in 2 for twice daily administration) administered orally for 7 days in Period 2 (14 days total treatment).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: PTC923 2.5 and 10 mg/kg/Day | Cohort 2: PTC923 5 and 20 mg/kg/Day | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.75 (5.123) | 11.55 (8.786) | 11.65 (6.659)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. TEAEs were defined as AEs that commenced or worsened after the first dose of study drug. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From first dose of study drug (Day 1) up to 30 (±3) days after last dose of study drug (up to 50 days)
Population: The Safety population included all randomized participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: PTC923 2.5 mg/kg/Day: Participants received PTC923 2.5 mg/kg/day for 7 days in Period 1.
- Cohort 1: PTC923 10 mg/kg/Day: Participants received PTC923 10 mg/kg/day for 7 days in Period 2.
- Cohort 2: PTC923 5 mg/kg/Day: Participants received PTC923 5 mg/kg/day for 7 days in Period 1.
- Cohort 2: PTC923 20 mg/kg/Day: Participants received PTC923 20 mg/kg/day for 7 days in Period 2.
Arm/Group | Cohort 1: PTC923 2.5 mg/kg/Day | Cohort 1: PTC923 10 mg/kg/Day | Cohort 2: PTC923 5 mg/kg/Day | Cohort 2: PTC923 20 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 4 | 4
Participants | 2 | 2 | 4 | 3

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PTC923 and Tetrahydrobiopterin (BH4)
Time Frame: Day 1 (pre-dose, within 30 minutes of dosing), 0.5, 1, 2, 4, 6, 8 hours postdose (prior to Day 1 evening dose), and 24 hours postdose (prior to Day 2 morning dose)
Population: The PK population included all participants who received at least 1 dose of study drug and had at least 1 quantifiable post-dose blood sample collected for analysis of PTC923, BH4, Phe, or Tyr concentrations. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | Cohort 1: PTC923 2.5 mg/kg/Day | Cohort 1: PTC923 10 mg/kg/Day | Cohort 2: PTC923 5 mg/kg/Day | Cohort 2: PTC923 20 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 3 | 3
nanograms (ng)/milliliter (mL)
  PTC923: number analyzed (Participants) | 0 | 4 | 3 | 3
  PTC923 |  | 1.110 (0.4031) | 0.533 (0.5033) | 2.120 (0.5292)
  BH4 | 19.455 (19.3731) | 109.375 (58.9440) | 48.200 (20.1570) | 275.030 (42.7941)

3. Secondary Outcome: Cmax of Phenylalanine (Phe) and Tyrosine (Tyr)
Time Frame: Day 1 (pre-dose, within 30 minutes of dosing), 0.5, 1, 2, 4, 6, 8 hours postdose (prior to Day 1 evening dose), 24 hours postdose (prior to Day 2 morning dose), 72 hours postdose (Day 4), on Day 7, and at the end of study (48 hours after last dose)
Population: The PK population included all participants who received at least 1 dose of study drug and had at least 1 quantifiable post-dose blood sample collected for analysis of PTC923, BH4, Phe, or Tyr concentrations. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micromoles (µmol)/liter (L)
Arm/Group | Cohort 1: PTC923 2.5 mg/kg/Day | Cohort 1: PTC923 10 mg/kg/Day | Cohort 2: PTC923 5 mg/kg/Day | Cohort 2: PTC923 20 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 3 | 3
micromoles (µmol)/liter (L)
  Phe | 939.35 (1059.225) | 725.98 (883.411) | 1420.30 (487.712) | 991.63 (555.802)
  Tyr | 157.15 (31.229) | 152.98 (22.314) | 173.40 (42.981) | 178.13 (48.925)

4. Secondary Outcome: Area Under the Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of PTC923 and BH4
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Cohort 1: PTC923 2.5 mg/kg/Day | Cohort 1: PTC923 10 mg/kg/Day | Cohort 2: PTC923 5 mg/kg/Day | Cohort 2: PTC923 20 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 3 | 3
hours*ng/mL
  PTC923: number analyzed (Participants) | 0 | 4 | 0 | 3
  PTC923 |  | 2.532 (2.2370) |  | 5.605 (1.0517)
  BH4 | 72.826 (62.8038) | 457.330 (204.2517) | 221.358 (82.6201) | 1158.337 (227.0332)

5. Secondary Outcome: AUC0-last of Phe and Tyr
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours*µmol/L
Arm/Group | Cohort 1: PTC923 2.5 mg/kg/Day | Cohort 1: PTC923 10 mg/kg/Day | Cohort 2: PTC923 5 mg/kg/Day | Cohort 2: PTC923 20 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 3 | 3
hours*µmol/L
  Phe | 3636.030 (4275.9593) | 1877.091 (1633.8636) | 3655.897 (1239.8499) | 2086.787 (871.7262)
  Tyr | 883.337 (65.2122) | 836.526 (143.4899) | 1037.085 (346.7325) | 1023.856 (368.7586)

6. Secondary Outcome: Time to Reach Cmax (Tmax) of PTC923 and BH4
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Groups:
- Cohort 2: PTC923 20 mg/kg/Day: Participants received 20 mg/kg/day for 7 days in Period 2.
Arm/Group | Cohort 1: PTC923 2.5 mg/kg/Day | Cohort 1: PTC923 10 mg/kg/Day | Cohort 2: PTC923 5 mg/kg/Day | Cohort 2: PTC923 20 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 3 | 3
hours
  PTC923: number analyzed (Participants) | 0 | 4 | 3 | 3
  PTC923 |  | 1.000 [0.50 to 2.03] | 1.000 [0.00 to 1.02] | 1.000 [0.98 to 2.00]
  BH4 | 4.017 [3.87 to 5.88] | 3.050 [2.00 to 4.05] | 4.000 [2.00 to 6.03] | 4.017 [2.00 to 4.05]

7. Secondary Outcome: Tmax of Phe and Tyr
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: PTC923 2.5 mg/kg/Day | Cohort 1: PTC923 10 mg/kg/Day | Cohort 2: PTC923 5 mg/kg/Day | Cohort 2: PTC923 20 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 3 | 3
hours
  Phe | 0.250 [0.00 to 0.50] | 0.517 [0.00 to 8.17] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  Tyr | 4.992 [3.87 to 7.37] | 4.025 [4.00 to 8.17] | 4.000 [4.00 to 7.03] | 2.000 [2.00 to 7.05]

8. Secondary Outcome: Change From Baseline (Day 1) in Plasma Phe Concentration at Day 7
Time Frame: Baseline (Day 1, pre-dose); Day 7
Population: The Efficacy population included all randomized participants who received any amount of study drug, and had available pre-dose Phe concentrations at Day 1 and at least 1 post-Day 1 visit within a given period. Here, 'Number analyzed' = participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Cohort 1: PTC923 2.5 mg/kg/Day | Cohort 1: PTC923 10 mg/kg/Day | Cohort 2: PTC923 5 mg/kg/Day | Cohort 2: PTC923 20 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 4 | 4
μmol/L
  Baseline | 884.20 (975.507) | 675.68 (842.579) | 1516.98 (442.673) | 971.48 (455.598)
  Change at Day 7: number analyzed (Participants) | 4 | 4 | 3 | 4
  Change at Day 7 | -812.25 (967.423) | -622.02 (840.853) | -1428.19 (531.327) | -913.63 (448.282)

9. Secondary Outcome: Number of Participants With Phe Concentrations in Acceptable Treatment Range of 130 to 360 μmol/L at Day 7
Time Frame: Day 7
Population: The Efficacy population included all randomized participants who received any amount of study drug, and had available pre-dose Phe concentrations at Day 1 and at least 1 post-Day 1 visit within a given period.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PTC923 2.5 mg/kg/Day | Cohort 1: PTC923 10 mg/kg/Day | Cohort 2: PTC923 5 mg/kg/Day | Cohort 2: PTC923 20 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 4 | 4
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Normal Blood Phe Concentrations <130 μmol/L at Day 7
Time Frame: Day 7
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PTC923 2.5 mg/kg/Day | Cohort 1: PTC923 10 mg/kg/Day | Cohort 2: PTC923 5 mg/kg/Day | Cohort 2: PTC923 20 mg/kg/Day
Number analyzed (Participants) | 4 | 4 | 4 | 4
Participants | 4 | 4 | 3 | 4

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) up to 30 (±3) days after last dose of study drug (up to 50 days)
Description: The Safety population included all randomized participants who received any amount of study drug.
Arm/Group | Cohort 1: PTC923 2.5 mg/kg/Day | Cohort 1: PTC923 10 mg/kg/Day | Cohort 2: PTC923 5 mg/kg/Day | Cohort 2: PTC923 20 mg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 2/4 | 4/4 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PTC923 2.5 mg/kg/Day (N=4) | Cohort 1: PTC923 10 mg/kg/Day (N=4) | Cohort 2: PTC923 5 mg/kg/Day (N=4) | Cohort 2: PTC923 20 mg/kg/Day (N=4)
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 1
Thirst (General disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Enuresis (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Eyelid infection (Infections and infestations) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT03519711/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT03519711/SAP_001.pdf